CLINICAL TRIAL: NCT01304017
Title: Virtual Reality Intervention for Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Dr. Harold Weingarden MD, Director of Day Rehabilitation Unit, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-10-8401-HW-CTIL
Record Dates: First submitted 2011-02-16; First posted 2011-02-25 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Stroke
Keywords: rehabilitation; stroke; intervention; physical activity; participation
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virtual Reality Therapy (Experimental): The VR-therapy will include the playing of various virtual reality or video-games which encourages the use of the extremities while sitting and standing.
  Interventions: Other: Virtual Reality
- Traditional Therapy (Active Comparator): The traditional therapy will include exercises for balance and walking and for the upper extremity using traditional therapeutic tools such as balls, weights, chairs, bands, steps, etc.
  Interventions: Other: Traditional Therapy

INTERVENTIONS:
Other: Virtual Reality — The VR-therapy will include the playing of various virtual reality or video-games which encourages the use of the extremities while sitting and standing
  Other Names: 'Community based' VR program
  Arms: Virtual Reality Therapy
Other: Traditional Therapy — The traditional therapy will include exercise for balance and walking and for the upper extremity using traditional therapeutic tools such as balls, weights, chairs, bands, steps, etc.
  Other Names: 'Community based' Traditional therapy program
  Arms: Traditional Therapy

SUMMARY:
In Israel approximately 16,000 people have a stroke each year. Most of these people suffer from weakness or paralysis of half of their body which leads to difficulties performing basic activities of daily life (BADL) such as dressing and walking. Due to the stroke, these individuals need to undergo intensive rehabilitation. After rehabilitation, physical activity has been strongly recommended to maintain their functional level which was achieved during rehabilitation. In addition regular physical activity can prevent secondary condition However, recent findings suggest that people with stroke do not perform enough physical activity with their upper and lower extremities.

The use of Virtual Reality (VR) for rehabilitation has been found to have potential for encouraging active purposeful movement. Many researchers have assessed the feasibility & usability of different VR systems and environments for individuals with stroke. Costly VR systems in addition to off-the-shelf video game consoles (e.g. Sony PlayStation EyeToy, Nintendo Wii) have been found to have great potential to encourage active purposeful movement. However, to date, only a limited number of studies have investigated the effectiveness of VR therapy post-stroke.

Since physical activity is important after stroke and the fact that individuals with stroke are not participating sufficiently in physical activity, I suggest to carry out this study.

The overall aim of this study is to assess the effectiveness of using novel technology of VR therapy to promote the participation in daily physical activity of individuals with stroke. A 'Community based' VR program will be compared to a traditional therapy program in promoting daily physical activity of the lower and upper extremities.

It is hypothesized that the VR intervention will be more efficient than the traditional therapy in promoting physical activity (walking and use of the weak upper extremity).

DETAILED DESCRIPTION:
In Israel there are approximately 16,000 new cases of stroke per year and recently stroke has been recognized by the Israeli health-care policy planners as a top priority disease. Individuals who have sustained a stroke constitute a large population with significant needs for rehabilitation. The most common symptom following stroke is paresis or paralysis to half of the body, contralateral to the side of brain lesion. These individuals experience difficulties performing basic activities of daily life (BADL) such as dressing and walking, in addition to instrumental activities of daily life (IADL) such as shopping and cooking.

Physical activity has been strongly recommended for these individuals to maintain their functional level which was achieved during rehabilitation. In addition regular physical activity can prevent secondary conditions such as heart disease, diabetes, obesity and decreases the risk of a recurrent stroke. Reduced physical activity can also lead to disuse atrophy and cardiovascular de-conditioning, which can result in deterioration of the person's physical condition. However, recent findings suggest that people with stroke do not perform enough physical activity with their upper and lower extremities.

The use of Virtual Reality (VR) for rehabilitation has been found to have potential for encouraging active purposeful movement. Many researchers have assessed the feasibility & usability of different VR systems and environments for individuals with stroke. Costly VR systems in addition to off-the-shelf video game consoles (e.g. Sony PlayStation EyeToy, Nintendo Wii) have been found to have great potential to encourage active purposeful movement. However, to date, only a limited number of studies have investigated the effectiveness of VR therapy post-stroke.

Since physical activity has been recognized to be a main factor in facilitating recovery post stroke and an important factor in preventing a recurrent stroke and due to the fact that individuals with stroke are not participating sufficiently in physical activity. Their physical and functional ability may deteriorate leading to expensive hospitalization and devastating outcomes, therefore, I suggest to carry out this study.

STUDY OBJECTIVES:

The overall aim of this study is to assess the effectiveness of using novel technology of VR therapy to promote the participation in daily physical activity of individuals with stroke. A 'Community based' VR program will be compared to a traditional therapy program in promoting daily physical activity of the lower and upper extremities.

METHODS:

A Randomized Controlled Trial (RCT) comparing VR therapy to traditional therapy will be applied. Eligible participants will be randomly allocated to the experimental or the control group. Blind assessors will assess their ability pre and post a 3-month intervention and at 3-month follow-up. Novel instrumentation of VR systems and video-game consoles will be applied for the intervention of the experimental group and accelerometers (that measure the intensity and duration of movement) will be utilized for assessing 'free-living' daily physical activity of the upper and lower extremities of both groups. In addition clinical assessments will be administered to assess the motor and functional ability of these individuals.

The main hypotheses are:

1. Daily walking post intervention will increase significantly more in the VR therapy groups compared to the traditional therapy groups.
2. Daily use of the weak upper extremity post intervention will increase significantly more in the VR therapy groups compared to the traditional therapy groups.
3. Daily walking on follow-up will be significantly higher in the VR therapy groups compared to the traditional therapy groups.
4. Daily use of the weak upper extremity on follow-up will increase significantly more in the VR therapy groups compared to the traditional therapy groups.

Secondary hypotheses;

1. Post intervention and on follow-up, the motor and functional ability of the weak upper extremity of the individuals in the VR therapy group will improve significantly more compared to the motor and functional ability of the weak upper extremity of individuals in the traditional therapy group.
2. Post intervention and on follow-up, the motor and functional ability of the weak lower extremity and balance of the individuals in the VR therapy group will improve significantly more compared to the individuals in the traditional therapy group.
3. Participation in ADL post intervention and on follow-up will be significantly higher in the VR therapy groups compared to the traditional therapy groups.
4. The executive functions of the individuals post intervention and on follow-up will be significantly higher in the VR therapy group compared to the traditional therapy group.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who have sustained a stroke at least 6 months prior to the study.
2. Are living in the community.
3. Are not receiving rehabilitation treatments.
4. Are experiencing difficulty using their legs and/or arms
5. Are able to walk 10 meters (with or without assistance)
6. Able to understand and follow simple instructions and to sign the informed consent form (assessed using MMSE score < 20/30 points).
7. Are willing to commit to attend two treatment sessions per week for 3 months.

Exclusion Criteria:

1. Have suffered in the past from epilepsy seizures
2. Have a neurological or orthopedic condition other than stroke that prevented independence in walking and BADL prior the stroke.
3. Have uncontrolled high blood pressure or unstable cardio-vascular condition (according to a letter from the family doctor).
4. Have vision deficits that cannot be corrected with glasses

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Physical activity of the lower and upper extremities | 6 months
  Physical activity of the lower and upper extremities will be measured using accelerometers to quantify the amount of hand usage, the number of steps taken per day and energy expenditure.

SECONDARY OUTCOMES:
The Fugl-Meyer Motor Assessment (FMA) (upper extremity subtest) | 6 months
  To assess the motor impairment of the upper extremity after stroke. Each movement is graded on a 3-point scale and the total score for the upper extremity ranges from 0-60 points.
The Action Research Arm Test (ARAT) | 6 months
  To assess the functional ability of the upper extremity by grasping and moving objects of different size and weight. It has four subtests; grasp, grip, pinch and gross movement. The total score is out of 57 points.
The Box and Blocks test | 6 months
  To assess manual dexterity. The subject is required to transfer as many blocks from one side of a box, over a divider, to the other side, in one minute. The number of blocks transported from one side of a box to the other in one minute is counted.
The 10-meter walk test (10MWT) | 6 months
  To assess gait speed. Subjects will be asked to walk along a 14-m walkway at their comfortable walking speed using their usual walking aids. Gait speed will be calculated from the time taken to traverse the middle 10 meters, as measured by a stop-watch. The average speed will be calculated from 3 trials.
Timed get up & Go Test | 6 months
  To measure mobility. It includes standing from a seating position, walking, turning, stopping, and sitting down which are all important tasks needed for a person to be independently mobile. For the test, the person is asked to stand up from a standard chair and walk a distance of 3 meters, turn around and walk back to the chair and sit down again. The time to complete this is recorded.
The Executive Functions Route Finding Test (EFRT) | 6 months
  To assess Executive Functioning. It involves the finding of an unfamiliar destination (office/room), located on a different floor from their current location. The examiner follows the participant and provides specific cues when needed.
Walking while Talking (WWT) | 6 months
  To assess the ability to divide and switch attention between 2 tasks during a 6 meter walk, turn and return. Subjects will walk while reciting consecutive letters of the alphabet aloud and while reciting alternate letters of the alphabet (i.e., a, c, e,…). The walking time and the number of mistakes will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Rand, PhD, Study Director — Tel Aviv University; Harold Weingarden, MD, Principal Investigator — Sheba Medical Center

REFERENCES:
- [Derived] Givon N, Zeilig G, Weingarden H, Rand D. Video-games used in a group setting is feasible and effective to improve indicators of physical activity in individuals with chronic stroke: a randomized controlled trial. Clin Rehabil. 2016 Apr;30(4):383-92. doi: 10.1177/0269215515584382. Epub 2015 May 7. PMID 25952586